CLINICAL TRIAL: NCT00936429
Title: Phase 1, Placebo-Controlled, Double-Blind, Safety Study of HBV-001 D1 in Healthy Adults
Brief Title: Study of HBV-001 D1 in Healthy Adults
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Hawaii Biotech, Inc. (Industry)
Responsible Party: Michele Yelmene, Hawaii Biotech, Inc
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: HBV-001-C-101
Record Dates: First submitted 2009-07-08; First posted 2009-07-10 (Estimated); Last update posted 2011-02-07 (Estimated); Status verified 2011-02

CONDITIONS: Dengue Fever
Keywords: Dengue fever; Dengue hemorrhagic fever; Dengue shock syndrome; Vaccine; Hawaii Biotech
MeSH Terms: conditions — Dengue; Severe Dengue | interventions — Aluminum Hydroxide

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- 10 µg DEN1-80E + 3.5 mg Alhydrogel (Experimental): Administration of 10 µg DEN1-80E vaccine at Weeks 0, 4, and 8.
  Interventions: Biological: DEN1-80E (HBV-001 D1 + 3.5 mg Alhydrogel)
- 50 µg DEN1-80E + 3.5 mg Alhydrogel (Experimental): Administration of 50 µg DEN1-80E vaccine at Weeks 0, 4, and 8.
  Interventions: Biological: DEN1-80E (HBV-001 D1 + 3.5 mg Alhydrogel)
- Placebo (Placebo Comparator): Administration of placebo vaccine at Weeks 0, 4, and 8.
  Interventions: Biological: Placebo for DEN1-80E

INTERVENTIONS:
Biological: DEN1-80E (HBV-001 D1 + 3.5 mg Alhydrogel) — 3 doses of DEN1-80E vaccine administered as 0.5 ml intramuscularly in deltoid.
  Other Names: HBV-001 D1
  Arms: 10 µg DEN1-80E + 3.5 mg Alhydrogel; 50 µg DEN1-80E + 3.5 mg Alhydrogel
Biological: Placebo for DEN1-80E — 3 doses of placebo vaccine administered as 0.5 ml intramuscularly in deltoid.
  Arms: Placebo

SUMMARY:
This is a single-center, double-blind, randomized, Phase 1 study to assess the safety and tolerability of HBV-001 D1 in healthy adult subjects.

DETAILED DESCRIPTION:
This is a single-center, double-blind, randomized, Phase 1 study to assess the safety and tolerability of HBV-001 D1 in healthy adult subjects. This will be an upward titration of two dose levels of HBV-001 D1 (10 µg and 50 µg of DEN1-80E) in 16 subjects across two cohorts. Participants in each cohort will receive HBV-001 D1 vaccine or placebo on Visits 1, 3 and 5.

ELIGIBILITY:
Inclusion Criteria:

* Males or females age 18 to 45.
* Body weight ≥ 110 pounds (50 kg).
* Satisfactory medical condition established by medical history and physical examination.
* Females must be of non-child bearing potential (i.e., surgically sterile) or, if of child-bearing potential must be abstinent or willing to employ adequate means of contraception.

Exclusion Criteria:

* Positive serum test for HIV, Hepatitis B surface antigens (HBsAg) and/or Hepatitis C antibodies.
* Abuse of drugs or alcohol within 12 months prior to screening.
* Use of corticosteroids or immunosuppressive drugs within 30 days of screening (use of topical or nasal corticosteroids is allowed).
* Any confirmed or suspected immunosuppressive or immunodeficient condition.
* Receipt of any vaccination within 30 days prior to screening.
* Receipt of blood products within 6 months of screening.
* Previous flavivirus vaccination (e.g., Japanese encephalitis or yellow fever) or flavivirus vaccination planned during the study period.
* History of flavivirus infection.
* No easy access to a fixed or mobile telephone.
* History of residing in a country endemic for dengue, Japanese encephalitis virus, or Yellow Fever virus for a period of > 1 year.
* Donation of ≥ 450 mL of blood within the previous 12 weeks.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2009-07; Primary Completion 2010-07 (Actual); Study Completion 2011-01 (Actual)

PRIMARY OUTCOMES:
To determine the safety of the study vaccine formulations in healthy adult subjects by assessing adverse events and laboratory data | Assessed at each study visit

SECONDARY OUTCOMES:
To assess the impact of vaccine dose level on immunogenicity determined by the levels of neutralizing antibodies and cell mediated immune responses | Every 2 weeks during treatment

CONTACTS AND LOCATIONS:
Overall Officials: Beth-Ann Coller, PhD, Study Director — Hawaii Biotech, Inc.
Locations (1):
- Saint Louis University, St Louis, Missouri, United States

REFERENCES:
- [Derived] Durbin AP, Pierce KK, Kirkpatrick BD, Grier P, Sabundayo BP, He H, Sausser M, Russell AF, Martin J, Hyatt D, Cook M, Sachs JR, Lee AW, Wang L, Coller BA, Whitehead SS. Immunogenicity and Safety of a Tetravalent Recombinant Subunit Dengue Vaccine in Adults Previously Vaccinated with a Live Attenuated Tetravalent Dengue Vaccine: Results of a Phase-I Randomized Clinical Trial. Am J Trop Med Hyg. 2020 Aug;103(2):855-863. doi: 10.4269/ajtmh.20-0042. Epub 2020 May 7. PMID 32394880
- [Derived] Manoff SB, George SL, Bett AJ, Yelmene ML, Dhanasekaran G, Eggemeyer L, Sausser ML, Dubey SA, Casimiro DR, Clements DE, Martyak T, Pai V, Parks DE, Coller BA. Preclinical and clinical development of a dengue recombinant subunit vaccine. Vaccine. 2015 Dec 10;33(50):7126-34. doi: 10.1016/j.vaccine.2015.09.101. Epub 2015 Oct 14. PMID 26458804